CLINICAL TRIAL: NCT05070754
Title: Using a Cold Atmospheric Plasma Device to Treat Molluscum Contagiosum and Verruca Vulgaris in Pediatric Patients
Brief Title: Cold Atmospheric Plasma Device for Pediatric Molluscum and Verruca
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: The Skin Center Dermatology Group (Industry)
Responsible Party: Principal Investigator, Lara Wine Lee, Assistant Professor, Dermatology and Dermatologic Surgery, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 106689
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Verruca Vulgaris; Molluscum Contagiosum Skin Infection
Keywords: Plasma; Cryotherapy; Pediatrics; Warts; Molluscum; Dermatology; Cantharidin
MeSH Terms: conditions — Warts | interventions — Cryotherapy; Cantharidin

STUDY DESIGN:
Intervention Model Description: During a clinical care visit, if a patient is eligible and agrees to participate, lesions will be selected by the dermatologist prior to procedure.The lesions will be marked randomly for a certain treatment regimen. The number of lesions treated will not exceed standard of care (SOC) recommendations. They will be determined by provider assessment and anatomical location. Participants with one lesion will receive either non-thermal atmospheric plasma (NTAP) or SOC. SOC is cryotherapy for warts and cantharidin for molluscum. Participants with greater than 2 lesions will receive equal treatment of NTAP and SOC. The number of lesions treated will be based off the providers assessment and anatomical location. Treatment of a single lesion or an odd number of multiple lesions will be based off a randomized list. All SOC lesions will be treated first to reduce the number of patients not wanting return to the more painful modality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Cold Atmospheric Plasma (CAP) (Experimental): We are proposing a clinical trial of a floating electrode-dielectric barrier device (FE-DBD), a Cold Atmospheric Plasma (CAP) device for the treatment of Verrucae Vulgaris and Molluscum Contagiosum. While novel to the medical field, and especially to dermatology, there are already a number of publications regarding its use on human skin in adults and children. CAP devices utilize noble gases (such as helium) to deliver plasma state matter to the skin. As its name implies, the generated plasma stream is of near skin temperature and it exists on normal atmospheric pressure. During the generation of the plasma there is no electric contact with the patient. The treatment does not increase skin surface temperature and the used helium gas, the same as used for balloons, being a noble gas does not cause a chemical reaction with the skin. The flow of the gas is slow, thus there is no mechanical effect on the skin.
  Interventions: Device: Floating electrode-dielectric barrier device (FE-DBD) cold atmospheric plasma (CAP)
- Cryotherapy (Active Comparator): Current standard of care (SOC) for treating Verruca Vulgaris in Children is cryotherapy. Patients randomized to this arm of the study will receive SOC treatment for their identified condition.
  Interventions: Device: Cryotherapy
- Cantharidin (Active Comparator): SOC for treatment of Molluscum Contagiosum is cantharidin. Patients randomized to this arm of the study will receive SOC treatment for their identified condition.
  Interventions: Drug: Canthardin Collodion

INTERVENTIONS:
Device: Floating electrode-dielectric barrier device (FE-DBD) cold atmospheric plasma (CAP) — The treatment device in this study generates cold atmospheric plasma. Cold atmospheric plasma has certain properties of plasma, such as ionized gas molecules. To create plasma, a pulse generator supplying 20 kilovolt pulse of 20-ns pulse width at 200 Hz (FPG10-01NM10, FID GmbH, Burbach, Germany) to a 5-mm diameter quartz-covered copper electrode of 10-cm length and 1 - 13mm quartz thickness. These nanosecond pulse parameters were chosen to provide sufficient treatment dose at the high level of plasma uniformity required to avoid any tissue damage. We will treat the lesions for approximately 1 to 2 minutes each, moving the electrode gently over the treatment area.
  Other Names: Non-thermal atmospheric pressure plasma (NTAP)
  Arms: Cold Atmospheric Plasma (CAP)
Device: Cryotherapy — Cryotherapy refers to the application of liquid nitrogen using a cryospray device in order to freeze a lesion of interest. Treatment is repeated every few weeks until the lesion of interest has disappeared. It is considered SOC for the treatment of warts.
  Other Names: Cold Therapy; Liquid Nitrogen
  Arms: Cryotherapy
Drug: Canthardin Collodion — Chemical compound that acts as a vesicant to form a blister around treatment area. The blister lifts the lesion of interest away from the skin, causing it to slough off in a few days. It is used as SOC for the treatment of Molluscum Contagiosum.
  Other Names: Cantharidin
  Arms: Cantharidin

SUMMARY:
This study is going to test a cold atmospheric plasma device (CAP), in particular a floating electrode-dielectric barrier device (FE-DBD), to treat warts and molluscum. The treatment device in this study generates cold atmospheric plasma (gaseous ionized molecules) to rid the virus from the body. Based on the successes of previous dermatologic studies, FE-DBD is being tested for this study to treat warts and molluscum. Patients will be enrolled to test the efficacy and safety of this device. The duration of the study is 4-12 weeks depending on treatment clearance. The number of lesions will be chosen by the dermatologist. Patients will receive standard of care therapy and/or NTAP depending on the number of lesions.

ELIGIBILITY:
Inclusion Criteria:

* All patients from 4-21 years old with at least 1 lesion of either verruca vulgaris or molluscum contagiosum
* Willingness of the participant and their guardian to provide consent when applicable

Exclusion Criteria:

* Unwillingness to participate in the study
* Received any treatment on the lesion in the past month, as determined by review of participant medical record
* Immunodeficiency as determined by review of participant medical record
* Adverse response to prior treatments as determined by review of medical record
* Signs of self-resolution as determined by study team members
* Conditions that lead to excessive scarring as determined by study team members
* Facial and genital lesions as determined by study team members

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Wine Lee, MD, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: lesions
Groups:
- Cold Atmospheric Plasma (CAP) Only: We conducted clinical trial of a floating electrode-dielectric barrier device (FE-DBD), a Cold Atmospheric Plasma (CAP) device for treatment of Verrucae Vulgaris and Molluscum Contagiosum. While novel to dermatology, publications exist regarding its use on human skin in adults and children. CAP devices utilize noble gases (such as helium) to deliver plasma state matter to the skin. The generated plasma stream is near skin temperature and exists on normal atmospheric pressure. In generation of plasma, there is no electric contact with the patient. Treatment does not increase skin surface temperature; the used helium gas is a noble gas and does not cause a chemical reaction with the skin. Flow of the gas is slow, thus there is no mechanical effect on skin.
  Floating electrode-dielectric barrier device (FE-DBD) cold atmospheric plasma (CAP): The treatment device in this study generates CAP. CAP has certain properties of plasma, such as ionized gas molecules. To create plasma, a pulse generator, which supplied 17 kHz, 6 µs width pulse at a power density of approximately 2 W/cm2 (AAPlasma, Philadelphia, PA) was connected to a 10 mm diameter quartz-covered copper electrode of 50 mm length and 1 mm quartz thickness with one end fused. These nanosecond pulse parameters were chosen to provide sufficient treatment dose at the high level of plasma uniformity required to avoid any tissue damage. We treated lesions for 2 minutes each, moving the electrode gently over the treatment area.
- Cryotherapy Only: Current standard of care (SOC) for treating Verruca Vulgaris in Children is cryotherapy. Patients randomized to this arm of the study have only one verruca lesion enrolled, and will receive SOC treatment for their identified condition.
  Cryotherapy: Cryotherapy refers to the application of liquid nitrogen using a cryospray device in order to freeze a lesion of interest. Treatment is repeated every few weeks until the lesion of interest has disappeared. It is considered SOC for the treatment of warts.
- CAP and Cryotherapy: Patients in this arm have more than one verruca lesion enrolled in the study. Thus, some of their lesions received CAP and some received SOC cryotherapy.
- CAP and Cantharidin: SOC for treatment of Molluscum Contagiosum is cantharidin. Patients randomized to this arm of the study will have multiple lesions, with some receiving cantharidin SOC treatment for their identified condition and some receiving cold atmospheric plasma (CAP).
  Canthardin Collodion: Chemical compound that acts as a vesicant to form a blister around treatment area. The blister lifts the lesion of interest away from the skin, causing it to slough off in a few days. It is used as SOC for the treatment of Molluscum Contagiosum.
Period: Overall Study
Arm/Group | Cold Atmospheric Plasma (CAP) Only | Cryotherapy Only | CAP and Cryotherapy | CAP and Cantharidin
Started (Patients could have up to 20 lesions enrolled. The lesions were randomized 1:1 to receive either CAP or standard of care therapy (cryotherapy for verruca or cantharidin for molluscum). Patients with only one lesion enrolled had that lesion randomized to either CAP or SOC.) | 2; 2 lesions | 1; 1 lesions | 11; 109 lesions | 3; 37 lesions
CAP | 2; 2 lesions | 0; 0 lesions | 11; 54 lesions | 3; 19 lesions
Cryotherapy | 0; 0 lesions | 1; 1 lesions | 11; 55 lesions | 0; 0 lesions
Cantharidin | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 3; 18 lesions
Completed | 2; 2 lesions | 1; 1 lesions | 11; 109 lesions | 1; 20 lesions
Not Completed | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 2; 17 lesions
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: Lesions
Groups:
- Total: Total of all reporting groups
Arm/Group | Cold Atmospheric Plasma (CAP) Only | Cryotherapy Only | CAP and Cryotherapy | CAP and Cantharidin | Total
Number analyzed (Participants) | 2 | 1 | 11 | 3 | 17
Number analyzed (Lesions) | 2 | 1 | 109 | 37 | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 11 | 3 | 17
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 6.5 [5 to 8] | 10 [10 to 10] | 10 [7 to 14] | 7 [4 to 13] | 9.1 [4 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 2 | 6
  Male | 1 | 0 | 9 | 1 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 2 | 1 | 10 | 2 | 15
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 11 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Lesions With no Response
Description: Absence of change in appearance of targeted lesion. Molluscum is defined as the visualization of a central umbilication with polylobular, white to yellow, amorphous structures. A peripheral crown of radiating or punctiform vessels may also be present. Warts are defined as grouped papillae, with dotted or loop vessels, and/or hemorrhagic points and lines often surrounded by a whitish halo.
Time Frame: 12 weeks
Population: The analyzed unit for this outcome is individual lesions. The sum of the number of participants in the two categories being higher than the total number of participants enrolled in the study is a result of the two categories not being mutually exclusive, as participants could have multiple lesions enrolled that were randomized to either CAP or SOC.
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Groups:
- Lesions Treated With Cold Atmospheric Plasma (CAP): This arm represents lesions that were randomized to receive treatment with cold atmospheric plasma (CAP) therapy.
- Lesions Treated With Standard of Care (SOC): This arm represents lesions that were randomized to receive SOC therapy (cryotherapy or cantharidin, depending on the lesion).
Arm/Group | Lesions Treated With Cold Atmospheric Plasma (CAP) | Lesions Treated With Standard of Care (SOC)
Number analyzed (Participants) | 16 | 15
Number analyzed (lesions) | 75 | 74
lesions | 8 | 9
Statistical Analysis 1: Comparison: Lesions Treated With Standard of Care (SOC); Outcome measures 1-3 were all tested together. Null hypothesis was that there was no difference in the degree of lesion resolution between the two treatment methods; Test type: Superiority; p = 0.534, Chi-squared

2. Primary Outcome: Numbers of Lesions With Partial Response
Description: There is change in the size, dyspigmentation, or discomfort of the targeted lesion as compared to its appearance and symptoms at the initial visit, but the lesion remains grossly visible. Molluscum is defined as the visualization of a central umbilication with polylobular, white to yellow, amorphous structures. A peripheral crown of radiating or punctiform vessels may also be present. Warts are defined as grouped papillae, with dotted or loop vessels, and/or hemorrhagic points and lines often surrounded by a whitish halo. Changes in the characteristics of the targeted lesions will be evaluated by a dermatologist and documented via photographs at follow-up visits at 4, 8, and 12 weeks, with the final outcome measured at the 12-week visit.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Lesions Treated With Cold Atmospheric Plasma (CAP) | Lesions Treated With Standard of Care (SOC)
Number analyzed (Participants) | 16 | 15
Number analyzed (lesions) | 75 | 74
lesions | 23 | 15
Statistical Analysis 1: Comparison: Lesions Treated With Standard of Care (SOC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.534, Chi-squared

3. Primary Outcome: Numbers of Lesions With Complete Response
Description: Targeted lesion is no longer grossly visible.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Lesions Treated With Cold Atmospheric Plasma (CAP) | Lesions Treated With Standard of Care (SOC)
Number analyzed (Participants) | 16 | 15
Number analyzed (lesions) | 75 | 74
lesions | 40 | 45
Statistical Analysis 1: Comparison: Lesions Treated With Standard of Care (SOC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.534, Chi-squared

4. Secondary Outcome: Post-Treatment CAP Tolerability Questionnaire
Description: This questionnaire measures tolerability of cold atmospheric plasma treatment. Assessment of dryness, peeling, scaling, erythema, edema, stinging, burning sensation, itching, scarring and dyspigmentation will each be assessed individually. Participants were asked about these symptoms at a 1-week post-first treatment phone call, and then at every in-person follow up visit. Outcome data represents the number of total lesions in each treatment group in which a participant reported at least one of the above adverse symptoms. Results of specific AEs are detailed in the Adverse Event section.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Lesions Treated With Cold Atmospheric Plasma (CAP) | Lesions Treated With Standard of Care (SOC)
Number analyzed (Participants) | 16 | 15
Number analyzed (lesions) | 75 | 74
lesions | 10 | 42
Statistical Analysis 1: Comparison: Lesions Treated With Standard of Care (SOC); Test type: Superiority; p < 0.001, Chi-squared

5. Secondary Outcome: Score of Visual Analogue Scale Associated With Treatment
Description: The visual analogue scale (VAS) is a validated subjective measurement of pain experienced by the patient. It consists of visual-numeric scale, numbered from 0-10. (0) indicate absence of pain or "no pain at all", while (10) indicates severe pain or "worst imaginable pain". This is supplemented by six faces with different expressions, ranging from happy to extremely upset. Each facial expression is assigned a numerical scale from 0 to 10.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: units from 0-10 on VAS scale
Units Other Than Participants: lesions
Arm/Group | Lesions Treated With Cold Atmospheric Plasma (CAP) | Lesions Treated With Standard of Care (SOC)
Number analyzed (Participants) | 16 | 15
Number analyzed (lesions) | 75 | 74
units from 0-10 on VAS scale | 2.5 [0 to 10] | 0.9 [0 to 8]
Statistical Analysis 1: Comparison: Lesions Treated With Standard of Care (SOC); Null hypothesis: there was no difference in median pain levels between SOC and NTAP treated lesions; Test type: Superiority; p = 0.142, Wilcoxon Signed Rank Test

ADVERSE EVENTS:
Time Frame: 4 months (maximum of 3 months of treatment, then 1 month post-treatment)
Description: Adverse events were categorized as patient-reported events or physician-determined sequelae post-treatment.
Arm/Group | Cold Atmospheric Plasma (CAP) Only | Cryotherapy Only | CAP and Cryotherapy | CAP and Cantharidin
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/11 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/11 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 9/11 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cold Atmospheric Plasma (CAP) Only (N=2) | Cryotherapy Only (N=1) | CAP and Cryotherapy (N=11) | CAP and Cantharidin (N=3)
Patient-reported AE: Pain (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0 — Patients reporting pain within individual lesions within 1 week of first treatment.
Patient-reported AE: Redness (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3
Patient-Reported AE: Other Color Change (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Patient-Reported AE: Blistering (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Patient-Reported AE: Scabbing (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Physician-determined Sequela: Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 8 | 3
Physician-determined Sequela: Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 6 | 2
Physician-determined Sequela: Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Physician-determined Sequela: Scarring (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
Limitations:

* Study was adequately powered with the number of lesions, but a small number of patients enrolled
* Low enrollment of patients with skin of color
* Patients limited to only three treatments with the NTAP device
* Assessment of sustained treatment response was limited to 4 weeks after treatment & may not represent long-term response
* Post-treatment sequelae were measured at the end of the study period. We are unable to determine whether they persisted or self-resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT05070754/Prot_SAP_000.pdf